CLINICAL TRIAL: NCT04852549
Title: Effects of Oculomotor Exercises on Balance, Dynamic Visual Acuity and Performance in Volleyball Players
Brief Title: Effects of Oculomotor Exercises on Volleyball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, elif yazgan, Principal investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Elif Aleyna Yazgan
Record Dates: First submitted 2021-04-08; First posted 2021-04-21 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Athlete
Keywords: Volleyball; Balance; Performance; visual acuity

STUDY DESIGN:
Intervention Model Description: The group of the cases meeting the criteria was determined by the numbers determined by the randomizer program in the "Research Randomiser" web site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No intervention group (No Intervention): The control group continued with routine training after evaluations.
- Oculomotor exercise group (Experimental): After the evaluation, the intervention group performed oculo-motor exercises for 4 weeks, 6 days a week, morning and evening, twice a day for 10 minutes, in addition to normal ball training. While doing the exercises, individuals were taught to focus on the purpose they held in their hands, move their head, and aim fast enough to see the image clearly. Two repetitions each week were added to the exercise numbers. Ten seconds rest between two sets and five seconds rest between movements.
  Interventions: Other: Oculomotor exercise

INTERVENTIONS:
Other: Oculomotor exercise — 1. While holding the head in the middle position, holding two colored objects in both hands, looking at the object in the right hand without turning the head, counting up to 10 and looking at the object in the left hand and counting up to 10,
  2. While holding a fixed head in the middle position and holding a colored object in the right hand, following the object with the eyes while moving the right hand from right to left without turning the head and returning,
  3. With the head fixed in the middle position, with the right hand on the left, eyes are fixed on the hand-held colored object and turn the head to the right and left.
  4. The head will be fixed in the middle position, the eyes will be fixed on the colored object held in the right or left hand and the arm and the head will be turned to opposite directions.
  Arms: Oculomotor exercise group

SUMMARY:
The researcher aimed to investigate the effects of oculo-motor exercises on dynamic visual acuity, balance and performance of volleyball players whose performance can be improved with visual skills training.

H0: Oculo-motor exercises applied to volleyball players are effective on dynamic visual acuity, balance and performance.

H1: Oculo-motor exercises have no effect on dynamic visual acuity, balance and performance in volleyball players.

DETAILED DESCRIPTION:
This study on the Effect of Oculo-Motor Exercises on Dynamic Visual Acuity, Balance and Performance in Volleyball Players was ethically approved by the "Istanbul Medipol University Non-Invasive Ethics Committee" with file number 10840098-604.01.01-E.14171 on 16.04.2020. The study included 52 female volleyball players aged 16-26 who played participants for at least 3 years without interruption. Power analysis was performed using the 3.1.9.5 version of the G-Power program to determine the number of individuals to be included in the study. Type-1 was accepted as 0.05 and power ratio as 80%. Effect size 0.8 was taken. According to the results of the power analysis, the number of participants required to be included in the study was determined as 52.

Participants; Age, height, weight, gender, body mass index, dominant side, position played in volleyball, number of weekly training, daily training time, previous sports injuries, education status, smoking and alcohol use, accompanying illnesses were questioned. FBT and YBT were used for balance evaluations, and Nelson's Hand Reaction Test was used for reaction times. In addition, Dynamic Visual Acuity and Vertical Jumping distances were evaluated twice before and after treatment.

Participants included in the study, the control group continued their routine ball training after the evaluations, while the intervention group continued with the oculo-motor training for 4 weeks, 6 days a week, in the morning and evening, for 10 minutes, 2 times a day, in addition to normal ball training. they did the exercises. While doing the exercises, individuals were taught to focus on the purpose they held in their hands, move their head, and aim fast enough to see the image clearly. Two repetitions each week were added to the exercise numbers. Ten seconds rest between two sets and five seconds rest between movements.

ELIGIBILITY:
Inclusion Criteria:

* Being in the age range of 16-26
* Playing licensed volleyball for at least 3 years without interruption
* Have normal vision and hearing

Exclusion Criteria:

* Having a direct blow to the lower or upper extremity in the past month
* People with musculoskeletal disorders may experience balance (forward head posture).
* Refractive defects
* History of ankle fracture
* Double-sided ankle sprain
* Vision problems
* History of lower extremity surgery in the last 6 months

Ages: 16 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-04-06 (Actual)

PRIMARY OUTCOMES:
Balance | The evaluation will be made after 4 weeks of training.
  Static balance of the individuals was evaluated by Flamingo Balance Test (FDT). A wooden stick of 50 cm length, 5 cm height and 3 cm width was used in the test. Dynamic balance changes of individuals were evaluated with YDT. In the measurement of dynamic balance with Y Balance Test (YDT), the amount of reaching out on the dominant sides of all individuals was measured.
Reaction time | The evaluation will be made after 4 weeks of training.
  Reaction time Nelson hand reaction test was used.
Dynamic visual acuity | The evaluation will be made after 4 weeks of training.
  In fact, dynamic vision is defined as the ability to detect details when there is a relative movement between the observer and the target object. It was measured by reading the numbers during neck rotation. A PowerPoint containing 10 slides, each of which randomly had 5 numbers, was used to measure dynamic vision (the size of all numbers was 12 to 20 at the center of the page). Each page had 5 numbers with the same font and each person evaluated 10 pages
Vertical jump | The evaluation will be made after 4 weeks of training.
  Vertical jump test was used.

CONTACTS AND LOCATIONS:
Overall Officials: Pınar Kaya Ciddi, Study Director — İstanbul Medipol University
Locations (1):
- Elif Aleyna Yazgan, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No